CLINICAL TRIAL: NCT06559163
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Obexelimab in Patients With Systemic Lupus Erythematosus
Brief Title: A Study of Obexelimab in Patients With Systemic Lupus Erythematosus
Acronym: SunStone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB012-02-001
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obexelimab (Experimental): Obexelimab will be administered as a subcutaneous injection for 24 weeks.
  Interventions: Drug: Obexelimab
- Placebo (Placebo Comparator): Placebo will be administered as a subcutaneous injection for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obexelimab — Obexelimab is a monoclonal antibody that simultaneously binds CD19 and FcyRllb, resulting in down regulation of B cell activity.
  Arms: Obexelimab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study aims to examine the efficacy and safety of obexelimab in participants with systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
This study consists of a 24-week treatment period followed by a 12-week follow-up period. Patients must have a clinical diagnosis of SLE at least 24 weeks prior to screening and meet the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) Classification Criteria. To enter the Screening Period (Day -28 to Day -1) patients will have active SLE as defined by having: a) hybrid Systemic Lupus Erythematosus Disease Activity Index (hSLEDAI) ≥ 6 and clinical hSLEDAI ≥ 4, and b) British Isles Lupus Assessment Group (BILAG)-2004 Grade A or B in ≥ 1 organ system. Patients must be treated with one or more of the following background nonbiologic lupus standard of care therapies: oral corticosteroid, antimalarial, and/or immunosuppressant.

On Day 1, patients will be randomized 1:1 to obexelimab or placebo subcutaneous (SC) injection once per week (QW) for 24 weeks. All patients will return to the study site for scheduled visits at Week 2, Week 4, and then every 4 weeks thereafter until study completion. During the study, patients will undergo assessments for efficacy, safety, PK, PD, and immunogenicity.

Including screening and follow-up, the maximum duration of participation in this study for an individual patient is approximately 40 weeks (i.e., up to a 28-day Screening Period, 24-week Treatment Period, and a 12-week follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥ 18 to ≤ 70 years of age
2. Diagnosed with SLE at least 24 weeks prior to screening and meets the 2019 EULAR/ACR classification criteria.
3. Patient has all 3 of the following based on features active on the day of the visits:

   1. hSLEDAI ≥ 6 and clinical hSLEDAI ≥ 4 at screening, and clinical hSLEDAI ≥ 4 at Day 1 Note: Clinical points exclude laboratory tests, except proteinuria.
   2. BILAG-2004 Grade A or B in ≥ 1 organ system at screening and Day 1.
   3. In the opinion of the investigator and the central adjudicator, there is sufficient disease activity to warrant enrollment into a clinical study with an investigational agent.
4. Patients must be treated with one or more of the following background nonbiologic lupus standard of care therapies: oral corticosteroid, antimalarial, and/or immunosuppressant.

Exclusion Criteria:

1. Active lupus nephritis for which, in the opinion of the investigator or the central adjudicator, current medications are insufficient for patient's safety or additional therapy that is not permitted in the protocol is needed.
2. A history of thrombosis or embolism in the previous 6 months before the Screening visit, or previous 12 months associated with antiphospholipid syndrome (APS) or another relevant hypercoagulable state.
3. Any active skin conditions other than cutaneous lupus erythematosus (CLE) that may interfere with the study assessment of CLE such as, but not limited to, psoriasis, dermatomyositis, and systemic sclerosis.
4. Active severe neuropsychiatric or central nervous system SLE.
5. Current inflammatory disease other than SLE (including, but not limited to, rheumatoid arthritis, psoriatic arthritis, spondyloarthropathy, reactive arthritis, scleroderma, dermatomyositis) that may interfere with the assessment of lupus signs and symptoms in the opinion of the investigator or central adjudicator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 24 weeks
  Proportion of patients who achieve a response according to the BILAG-Based Composite Lupus Assessment (BICLA) Response

SECONDARY OUTCOMES:
Secondary Outcome Measures | 24 weeks
  Proportion of patients who achieve response according to the Systemic Lupus Erythematosus Responder Index 4 (SRI-4).

OTHER OUTCOMES:
Additional Outcome Measures | 24 weeks
  Number of patients with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and injection site reactions.

CONTACTS AND LOCATIONS:
Locations (81):
- United States (16):
  - Sierra Pacific Arthritis and Rheumatology Centers, Fresno, California
  - California Research Institute, Huntington Park, California
  - University of California, San Diego, La Jolla, California
  - Clinical Research of West Florida, Inc, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Accurate Clinical Research, Lake Charles, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - June DO, PC, Lansing, Michigan
  - Juno DO, PC, Lansing, Michigan
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Penn State - Hershey Medical Center, Hershey, Pennsylvania
  - Prolato Clinical Research Center (PCRC), Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Prime Clinical Research - Mansfield, Mansfield, Texas
- CHU de Liege, Liège, Belgium
- Bulgaria (2):
  - Medical Center Medtech Services EOOD, Haskovo
  - University Multiprofile Hospital for Active Treatment "Eurohospital Plovdiv", Plovdiv
- Canada (2):
  - Richmond Clinical Trials, Richmond, British Columbia
  - Riverside Professional Centre, Sydney, Nova Scotia
- China (12):
  - Anhui Provincial Hospital (The First Affiliated Hospital of USTC), Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangx
  - Lanzhou University Second Hospital, Pudong, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - The First Affiliated Hospital of Ziamen University, Xiamen
- Sjaellands Universitetshospital, Koge, Køge, Denmark
- Germany (2):
  - Medicover Munchen Ost MVZ, München, Bavaria
  - Uniklinik Koln, Cologne
- Greece (6):
  - Attikon University General Hospital, Chaïdári, Athens
  - General Hospital Asklepieio Voulas, Voula, Athens
  - University General Hospital of Heraklion, Heraklion
  - Olympion General Clinic, Pátrai
  - Kianous Stavros, Thessaloniki
  - General Hospital of Thessaloniki ''Hippokration'', Thessaloniki
- Italy (2):
  - Policlinico Universitario Campus Biomedico Di Roma, Roma
  - Centro Ricerche Cliniche Di Verona S.r.l., Verona
- Japan (5):
  - Hospital of Japan Community Health Care Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Hospital of Shinkenko Clinic, Naha, Okinawa
  - Hokkaido University Hospital, Kita-ku, Sapporo Hokkaido
  - Juntendo University Hospital, Bunkyō City
- Mexico (5):
  - Clinstile, S.A. de C.V., Mexico City, Cuidad de Mexico
  - PanAmerican Clinical Research, Guadalajara, Jalisco
  - Eme Red Hospitalaria, Mérida, Yucatán
  - Kohler and Milsten Research, Mérida, Yucatán
  - Oaxaca Site Management Organization, Oaxaca City
- Poland (8):
  - Prywatna Praktyka Lekarska Prof Hab Med Pawel Hrycaj, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Krakowskie Centrum Medyczne, Krakow
  - SOMED CR, Lodz
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Pracownia Badan Klinicznych Salus, Wroclaw
- Portugal (3):
  - Hospital Egas Moniz, Lisbon
  - ULS de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - ULS da Arrábida, E.P.E. - Hospital de São Bernardo, Setúbal
- Puerto Rico (2):
  - Centro Reumatologico de Caguas, Caguas, Puerto Rico
  - Latin Clinical Trial Center, San Juan, Puerto Rico
- Romania (2):
  - Centrul Medical de Diagnostic si Tratament Ambulator NEOMED SRL, Brasov
  - Dr I Cantacuzino Clinical Hospital, Bucharest
- South Africa (2):
  - FARMOVS, Bloemfontein
  - Panorama Medical Centre, Cape Town
- Spain (4):
  - FutureMeds DKF, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Taiwan (6):
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District